CLINICAL TRIAL: NCT03590639
Title: IBD-Disk Validation Study for Disability Assessment Functional of Patients With Inflammatory Diseases Intestinal Chronic
Brief Title: Validation Study for Disability Assessment Functional of Patients With Inflammatory Diseases Intestinal Chronic (VALIDate)
Acronym: VALIDate
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Angers (Other Government); Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC18_0032
Record Dates: First submitted 2018-06-08; First posted 2018-07-18 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2018-06

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Inflammatory Bowel Diseases; disability; quality of life; IBD Disk; IBD-Disability Index; Patient-Reported Outcomes
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory Bowel Diseases (IBD) often affect psychological, family, social and professional dimensions of patients' life, leading to disability which is essential to quantify as part of Patient-Reported Outcomes (PROs) newly included in the therapeutic targets to reach in IBD patients. Up to now, the IBD-Disability Index (IBD-DI) was the only validated tool to assess functional status, but it is not appropriate for use in clinical practice. The IBD Disk was then developed, a shortened and self-administered tool, adapted from the IBD-DI, in order to give immediate representation of patient-reported disability. However, the IBD Disk has not been validated yet in clinical practice. The aims of the VALIDate study is to validate this tool in a large population of French IBD patients and to compare it to the already validated IBD-DI.

DETAILED DESCRIPTION:
The IBD-Disk has not been evaluated in clinical practice and has not yet been validated. but the interest of rapid assessment of the disease led the physicians in University Hospital of Nantes' department, some of whom had participated in the construction of this tool, to use it in routine practice for consultations of patients with IBD, joined by many gastroenterologists from other hospitals including the University Hospitals of Rennes and Angers.

The objective of this study is to validate this tool and prove its effectiveness by comparing it to the gold standard represented by the IBD-DI, in the same way that the PsoDisk has been validated prospectively compared to other tools for evaluating the quality of life and activity of psoriatic disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes
* aged over 18 with an established diagnosis of IBD (Crohn's Disease, Ulcerative Colitis or IBD unclassified)

Exclusion Criteria:

* ongoing pregnancy or breast feeding woman
* vulnerable people i.e. Adults under a legal protection regime (guardianship, trusteeship, judicial safeguard )
* insufficient command of French language and relevant psychiatric comorbidities (both of them making the self-questionnaire difficult to fill in)
* uncertain IBD diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in 3 university hospitals (Nantes, Rennes, Angers) which use the IBD-Disk in their current practice.
  Investigators will offer patients with chronic inflammatory disease intestinal tract and seen in gastroenterological consultation during a control visit of their pathology to enter the study, regardless of previous or current treatments, with a goal to include 400 patients
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2020-04-16 (Actual)

PRIMARY OUTCOMES:
IBD Disk's validity | changes from baseline IBD disk at 12 months
  Validity of the questionnaire

SECONDARY OUTCOMES:
IBD Disk's reliability | Baseline and follow-up visit (between 3 and 12 months after baseline) for all of the outcome measures, except for reproducibility (7 days after baseline)
  IBD Disk's reliability (Cronbach's coefficient alpha)
IBD Disk's reproducibility | Baseline and follow-up visit (between 3 and 12 months after baseline) for all of the outcome measures, except for reproducibility (7 days after baseline)
  IBD Disk's reproducibility (test-retest reliability)
Satisfaction of the physician by Visual analog Scale | Baseline and follow-up visit (between 3 and 12 months after baseline) for all of the outcome measures, except for reproducibility (7 days after baseline)
  IBD Disk's feasibility (visual analog scale filled by the physician at the end of the study)
Correlation between the IBD-Disk and the seriousness of the pathology | Baseline and follow-up visit (between 3 and 12 months after baseline) for all of the outcome measures, except for reproducibility (7 days after baseline)
  the IBD-disk will be combined to the seriousness of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline TRANG, PH, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - Angers University Hospital, Angers
  - Nantes University Hospital, Nantes
  - Rennes University Hospital, Rennes

REFERENCES:
- [Derived] Le Berre C, Bourreille A, Flamant M, Bouguen G, Siproudhis L, Dewitte M, Dib N, Cesbron-Metivier E, Goronflot T, Hanf M, Gourraud PA, Kerdreux E, Poinas A, Trang-Poisson C. Protocol of a multicentric prospective cohort study for the VALIDation of the IBD-disk instrument for assessing disability in inflammatory bowel diseases: the VALIDate study. BMC Gastroenterol. 2020 Apr 16;20(1):110. doi: 10.1186/s12876-020-01246-7. PMID 32299390